CLINICAL TRIAL: NCT02294578
Title: Prospective Blinded Evaluation of Salivary Transcriptome Biomarkers for Non-small Cell Lung Cancer Detection
Brief Title: Salivary Biomarkers for Non-small Cell Lung Cancer Detection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PeriRx (Industry)
Responsible Party: Principal Investigator, Jack Martin, MD, Chief Medical Officer, PeriRx
Other Study IDs: PeriRx LC
Record Dates: First submitted 2014-11-05; First posted 2014-11-19 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer
Keywords: Biomarkers; saliva; mRNA
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lung Cancer: Patients with biopsy proven lung cancer
- Controls: Patients with lung lesions suspicious for the presence of cancer and with cancer excluded after further diagnostic study

SUMMARY:
The investigators plan to recruit patients for a prospective study in patients in need of evaluation for lung lesions suspicious for cancer. Saliva samples will be collected before diagnostic evaluation including biopsy with subsequent blinded examination of the salivary markers without knowledge of the disease status. This prospective recruitment with retrospective blinded evaluation or PRoBE design satisfies the highest standards recommended by the National Cancer Institute for biomarker development. This process limits the selection bias that can confound retrospective studies. As the primary endpoint, a pre-specified multi-marker panel will be evaluated based on the combination of sensitivity and specificity. In addition, seven pre-specified individual candidate mRNA cancer markers and six internal reference or "housekeeping" genes will be evaluated. The performance of new multi-marker panels will also be assessed and compared with the prior pre-specified model based on sensitivity and specificity combinations as well as the area under the receiver operating characteristic curve.

DETAILED DESCRIPTION:
Consecutive eligible patients presenting to the study institutions and associated clinics will be enrolled. Inclusion and exclusion criteria are detailed separately in the section on eligibility. The target enrollment population listed in the study design section provides a greater than 85% power to achieve the pre-specified goal for the sensitivity and specificity of the pre-specified model. Saliva will be collected in vials pre filled with mRNA stabilizer. Seven mRNA biomarkers (BRAF, CCNI, EGRF, FGF19, FRS2, GREB1, and LZTS1) will be measured in a central laboratory by quantitative PCR with the laboratory personnel blinded to the patient diagnosis. The primary outcome is the validation of a pre-specified multi-marker model. This pre-specified model incorporates 3 of the cancer genes and the housekeeping gene. The model will be validated based on the sum of sensitivity and specificity exceeding 1.3 with the lower limit of the 95% confidence interval exceeding 1.0. A secondary endpoint is the development of new multi-maker models with potential improved performance. These new models will be developed by logistic regression and compared with the pre-specified model based on the area under the receiver operating characteristic curve and the maximum sum of sensitivity and specificity. Individual candidate biomarkers will also be validated based on a statistically significant up-regulation in cancer patients compared with controls. Potential new housekeeping genes will be evaluated based on their equivalence in cancer and control as well as their performance in multi-marker models in comparison with the pre-specified housekeeping gene which is GADPH..

ELIGIBILITY:
Inclusion Criteria:

* Any patient presenting to the participating institutions of affiliated clinics for evaluation or biopsy of a lung lesion suspicious for cancer.
* Patients ≥ 18 years of age
* Patients willing and able to give informed consent

Exclusion Criteria:

* Diagnosis of cancer within the last two years, excluding non-melanoma skin cancer (if > 2 years since diagnosis, must be free of known disease & not on current treatment for cancer).
* Prior immunosuppressive therapy or autoimmune disorder
* Known HIV infection
* Known Hepatitis infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting for evaluation of lung lesions suspicious for the presence of lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Performance of a pre-specified multi-marker panel (incorporating 3 of the 7 pre-specified cancer genes and the housekeeping gene) | Patients will be followed until their work up determines if they have benign pathology or lung cancer and the stage is determined. The complete analysis of biomarkers will occur at approximately 15 months after the start of enrollment.
  Multi-marker test score conmined sensitivity abd specificity

SECONDARY OUTCOMES:
Validation of the individual mRNA biomarkers (BRAF, CCN1, EGRF, FGF19, FRS2,GREB1 and LZTS1) | Patients will be followed until their work up determines if they have benign pathology or lung cancer and the stage is determined. The complete analysis of biomarkers will occur at approximately 15 months after the start of enrollment.
  Delta Ct values based on PCR analysis comparing cancer and controls
Performance of new multi-marker models | Patients will be followed until their work up determines if they have benign pathology or lung cancer and the stage is determined. The complete analysis of biomarkers will occur at approximately 15 months after the start of enrollment.
  Multi-marker test score combined sensitivity and specificity
Performance of new candidate housekeeping genes | Patients will be followed until their work up determines if they have benign pathology or lung cancer and the stage is determined. The complete analysis of biomarkers will occur at approximately 15 months after the start of enrollment.
  Based on Normfinder stability

CONTACTS AND LOCATIONS:
Overall Officials: Jack L Martin, MD, Study Chair — PeriRx, LLC
Locations (2):
- United States (2):
  - St. John Macomb-Oakland Hospital, Warren, Michigan
  - Main Line Health Ststem, Wynnewood, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided